CLINICAL TRIAL: NCT01408849
Title: Use of Maytenus Ilicifolia Mart. ex Reiss in the Treatment of Dyspepsia
Brief Title: Use of Maytenus Ilicifolia in the Treatment of Dyspepsia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of adherence and huge loss of follow up.
Sponsor: Casa Espirita Terra de Ismael (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Fabio Carmona, Assistant Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Maytenus2011
Record Dates: First submitted 2011-07-29; First posted 2011-08-03 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Dyspepsia
Keywords: Endoscopy; Herbal medicine; Phytotherapy
MeSH Terms: conditions — Dyspepsia | interventions — Omeprazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Maytenus (Experimental): Tea of Martens ilicifolia leaves
  Interventions: Drug: Maytenus ilicifolia leaves infusion
- Omeprazole (Active Comparator): Omeprazole as active comparator
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: Maytenus ilicifolia leaves infusion — 2 g of powdered leaves in 150 mL of boiling water, 3 times a day, for 8 weeks
  Arms: Maytenus
Drug: Omeprazole — Standard therapy
  Arms: Omeprazole

SUMMARY:
This study aims to evaluate the therapeutic effect of the infusion of Maytenus ilicifolia Mart. ex Reiss leaves, used for 8 weeks, on patients with dyspepsia. Primary endpoint is SODA score, secondary endpoint is endoscopic classification (Sydney).

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* being literate
* diagnosis of dyspepsia
* initial SODA score > or = 25

Exclusion Criteria:

* pregnancy
* lactation
* allergy to Maytenus species
* fail to use the drug for 3 uninterrupted weeks
* new onset serious adverse events, attributable to the drug
* patient's request

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
SODA score | 8 weeks

SECONDARY OUTCOMES:
Sydney classification | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ana MS Pereira, PhD, Study Director — University of Ribeirao Preto; Jose S Santos, MD, PhD, Study Chair — HCFMRP-USP; Fabio Carmona, MD, PhD, Principal Investigator — HCFMRP-USP; Suzeidi B Castanheira, MD, PhD, Principal Investigator — HCFMRP-USP
Locations (1):
- Hospital das Clinicas FMRP-USP, Ribeirão Preto, São Paulo, Brazil